CLINICAL TRIAL: NCT02457130
Title: Comparison of TIcagrelor and Clopidogrel in Patients With Coronary Artery diseaSe and Type 2 Diabetes Mellitus (TICS-DM): a Randomized Pharmacodynamic Study
Brief Title: Comparison of TIcagrelor and Clopidogrel in Patients With Coronary Artery diseaSe and Type 2 Diabetes Mellitus (TICS-DM)
Acronym: TICS-DM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Spanish Society of Cardiology (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, José Luis Ferreiro, MD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0162
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus. Type 2
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): After providing written informed consent, eligible subjects will be randomized in a 1:1 fashion to group A or B.
  Ticagrelor (180-mg loading dose the first day followed by 90-mg b.i.d. maintenance dose) for one week; washout period of 2-4 weeks; crossover to clopidogrel (600-mg loading dose the first day followed by 75-mg daily maintenance dose) for one-week.
  Interventions: Drug: Ticagrelor; Drug: Clopidogrel
- Group B (Experimental): After providing written informed consent, eligible subjects will be randomized in a 1:1 fashion to group A or B.
  Clopidogrel (600-mg loading dose the first day followed by 75-mg daily maintenance dose) for one-week; washout period of 2-4 weeks; crossover to ticagrelor (180-mg loading dose the first day followed by 90-mg b.i.d. maintenance dose) for one week.
  Interventions: Drug: Ticagrelor; Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor
  Other Names: Brilinta
Drug: Clopidogrel
  Other Names: Plavix

SUMMARY:
Patients with type 2 diabetes mellitus (T2DM), have a high prevalence of suboptimal response to clopidogrel (up to 40%). This impaired response to antiplatelet drugs has been consistently associated with a higher risk of adverse ischemic outcomes. Different strategies have been suggested to overcome variability in response to clopidogrel and improve clinical outcomes in diabetic patients. One of these strategies is the use of newer P2Y12 inhibitors, such as ticagrelor, with more potent and consistent platelet inhibitory effects compared to clopidogrel. In summary, since patients with T2DM continue to have enhanced platelet reactivity despite the administration of commonly used dual antiplatelet therapy with aspirin and standard doses of clopidogrel, newer and more potent antiplatelet treatment strategies are warranted in this high-risk population. The purpose of the present study is to compare platelet inhibitory effects achieved with ticagrelor versus clopidogrel, both on top of aspirin therapy, in patients with type 2 DM and stable coronary artery disease.

DETAILED DESCRIPTION:
Despite the clinical benefit associated with dual therapy consisting in aspirin and clopidogrel, there are still a considerable number of patients who continue to have atherothrombotic events. Several studies have shown a wide interindividual variability in response to clopidogrel treatment and patients with poor response have an increased risk of recurrent ischemic events. In particular, patients with type 2 diabetes mellitus (T2DM), have a high prevalence of suboptimal response to clopidogrel (up to 40%). This impaired response to antiplatelet drugs has been consistently associated with a higher risk of adverse ischemic outcomes. Different strategies have been suggested to overcome variability in response to clopidogrel and improve clinical outcomes in diabetic patients. One of these strategies is the use of newer P2Y12 inhibitors, such as ticagrelor, with more potent and consistent platelet inhibitory effects compared to clopidogrel. In summary, since patients with T2DM continue to have enhanced platelet reactivity despite the administration of commonly used dual antiplatelet therapy with aspirin and standard doses of clopidogrel, newer and more potent antiplatelet treatment strategies are warranted in this high-risk population. The purpose of the present study is to compare platelet inhibitory effects achieved with ticagrelor versus clopidogrel, both on top of aspirin therapy, in patients with type 2 DM and stable coronary artery disease (CAD).

This is a multi-center prospective, open-label, two-sequence, two-period, randomized crossover study conducted in T2DM patients between the ages of 18 and 75 years with known CAD. Subjects will be randomized in a 1:1 fashion to take ticagrelor (180-mg loading dose the first day followed by 90-mg maintenance dose) or clopidogrel (600-mg loading dose the first day followed by 75-mg daily maintenance dose) for one-week on a background of aspirin therapy (100 mg daily). After a 2-4 week washout period, subjects will cross-over treatment regimen. The washout periods are included to minimize carryover effects between treatment regimens. Patient compliance will be assessed by interview and pill counting.

Platelet function testing will be performed at the following time-points (repeated in the two periods of treatment): baseline, 2 and 24 hours after taking loading dose of the assigned drug, and 1 week after initiating the assigned drug.

All statistical comparisons of platelet function for the primary and secondary endpoints will be conducted using linear mixed-effect models with treatment, sequence, period and treatment*period (treatment by period interaction in order to test for carryover effects) as fixed effects, subject as a random effect and baseline value of the corresponding platelet function test as a covariate. A two-tailed p value of less than 0.05 will be considered to indicate a statistically significant difference for all the analyses performed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Age between 18 and 75 years
* Type 2 DM according to ADA criteria
* Angiographically documented CAD
* Chronic treatment (>1 month) with aspirin (100mg/day)

Exclusion Criteria:

* Known allergies to aspirin, clopidogrel, or ticagrelor
* Blood dyscrasia
* Any recent acute coronary syndrome (<30 days) or hemodinamic instability
* Recent antiplatelet therapy (<14 days), with the exception of ASA, including: thienopyridines, cilostazol, dipiridamol, glycoprotein IIb/IIIa inhibitors
* Oral anticoagulation with a coumarin derivative
* Concomitant treatment with a potent CYP3A4 inhibitor (e.g. ketoconazole, claritromicine, nefazodone, ritonavir, atazanavir)
* Any active bleeding
* Recent history of stroke, TIA or intracranial bleeding (<6 months prior to inclusion)
* Platelet count <100x106/microl
* Severe chronic kidney disease (creatinine clearance measured with Cockcroft-Gault formula <30ml/min)
* Any active neoplasm
* Baseline ALT >2.5 times the upper limit of normality
* Pregnant or childbearing females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity | 7 days
  maximal platelet aggregation, measured with light transmittance aggregometry (using 20 μM ADP as agonist), achieved after 1 week of treatment with ticagrelor or clopidogrel

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Ferreiro, Principal Investigator — Hospital Universitari de Bellvitge - IDIBELL
Locations (3):
- Spain (3):
  - Hospital Universitari de Bellvitge - IDIBELL, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Murcia

REFERENCES:
- [Derived] Marcano AL, Gracida M, Roura G, Gomez-Lara J, Romaguera R, Teruel L, Fuentes L, Muntane-Carol G, Merono O, Sosa SG, Gomez-Hospital JA, Comin-Colet J, Ferreiro JL. Antiplatelet efficacy of ticagrelor versus clopidogrel in Mediterranean patients with diabetes mellitus and chronic coronary syndromes: A crossover pharmacodynamic investigation. Front Cardiovasc Med. 2022 Nov 22;9:1057331. doi: 10.3389/fcvm.2022.1057331. eCollection 2022. PMID 36483622